CLINICAL TRIAL: NCT02453178
Title: Effects of a Bicycling Intervention on Cognitive Skills and Cardiovascular Health
Acronym: BIKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Michelle W. Voss, Assistant Professor of Psychological and Brain Sciences, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201405837
Record Dates: First submitted 2015-04-25; First posted 2015-05-25 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Sedentary Lifestyle
Keywords: physical activity; aging; cognition; brain; exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steady state moderate intensity cycling (Experimental): Moderate intensity exercise training will be a 12-week supervised cycling program, with supervision directly from our research team. All participants will first receive a one-on-one orientation with an exercise training specialist that has been trained by Dr. Gary Pierce in monitoring an exercise program for healthy older adults. Training will start with a 5 minute-warm-up, 20 minutes moderate intensity cycling and 30 minutes passive cycling, and 5 minute cool-down per session, for 3 sessions/week. In each additional week, we will add 6 minutes of moderate intensity cycling per session, until the total time for moderate intensity is 50 minutes per session by the start of week 5 (with additional 5 minute warm-up and 5 minute cool-down).
  Interventions: Behavioral: Cycling
- Intermittent cycling (Active Comparator): The intermittent cycling group will come to the exercise lab for the same duration and frequency each week and complete primarily passive cycling such that a motor in the stationary bicycle moves the pedals for them. To maintain interest in this intervention, we will include short bouts of moderate intensity activity. The short bouts of moderate intensity cycling will be designed to be ineffective for substantially increasing cardiorespiratory fitness over the course of the intervention.
  Interventions: Behavioral: Cycling

INTERVENTIONS:
Behavioral: Cycling — The experimental group will complete a 3 month exercise program that includes working up to cycling at a moderate intensity for 50 minutes/session 3 times a week. The comparison group will complete a 3-month exercise program that includes intermittent cycling (alternating between passive and moderate intensity) for 50 minutes/session 3 times a week. Both groups will exercise in our laboratory at Spence Labs, and will be supervised by an exercise trainer that is trained in working with elderly and special populations.
  Other Names: Exercise

SUMMARY:
Although exercise is known to delay cognitive decline and decrease our risk of Alzheimer's Disease, there is a lack of understanding of how exercise protects the aging brain. The proposed research takes a novel approach to this problem by testing the concept that there are acute, direct effects of exercise in the same brain regions that are affected by chronic exercise training. If the investigators are successful, the acute paradigm will allow us to determine the critical exercise parameters that modulate brain function in humans using only a single exercise dose.

DETAILED DESCRIPTION:
Given the rising proportion of older adults worldwide and the progressive decline in brain function with advancing age, there is a pressing need to develop novel interventions that protect the aging brain. The predominant approach for implementing exercise training to improve brain function is to increase cardiovascular fitness. However, there is mixed empirical support for the effectiveness of this approach. Further, there are also acute effects of exercise within one hour of the cessation of a single exercise session. These effects occur before adaptations related to fitness could occur and animal studies have shown they occur in the same brain regions that benefit from longer-term exercise training. Therefore, the investigators propose the acute paradigm is a tool to probe this early, direct response from exercise in order to determine how best to maximize the long-term benefit of exercise training on the aging brain. This presents a critical need to determine the mechanistic relation between acute and long-term effects of exercise on the aging brain. Our long-term goal is to determine how exercise protects the brain from the adverse effects of aging. In turn, our specific objective in this R21 proposal is to support or refute the concept that a single session of exercise produces acute increases in functional synchrony of clinically relevant brain networks that are related to accrued exercise-training effects in the same brain systems. Our central hypothesis is that the effects of moderate intensity exercise will increase the functional synchrony of the hippocampus with the Default Mode Network, and the Prefrontal Cortex with the Fronto-Executive Network, in the same fashion as a 12-week moderate intensity exercise training program. This hypothesis is based on data showing acute effects of exercise on factors related to neuronal plasticity and excitability in the same brain regions that show long-term effects of exercise in animals. The contribution of the proposed research is significant because it will determine the extent to which the acute exercise paradigm can provide insight into how regular exercise protects the brain from adverse effects of aging. The proposed research is innovative because for the first time the investigators will examine the overlapping neural systems and outcomes associated with acute and chronic exercise in the same individuals. Overall, success in this project will enable future research to study how varying exercise parameters such as mode or intensity affect exercise-induced change in brain function and the timecourse of these effects, as well as the neurobiological mechanisms associated with the direct effects of exercise on the aging brain.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to participate in an aerobic exercise intervention based on the Physical Activity Readiness Questionnaire, and corrected vision of 20/40.
* Because our older adult sample is over the age of 40, we will also require completion of a detailed health history questionnaire and further eligibility for the exercise intervention will be determined following approval from a physician that monitored electrocardiography (ECG) response during a maximal aerobic fitness test that is part of the second study visit described below.

Exclusion Criteria:

* Not between the ages of 60 and 80 years old
* Not fluent in English
* Score < 26 (out of 30) on the Montreal Cognitive Assessment (MoCA)
* Inability to comply with experimental instructions
* Qualify as "high risk" for acute cardiovascular event by the published standards of the American College of Sports Medicine
* Left-handed
* Previous diagnosis of neurological, metabolic, or psychiatric condition, and no previous brain injury associated with loss of consciousness
* Inability to complete an MRI

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Functional brain network integrity: the strength of the correlation between fluctuating functional magnetic resonance imaging (fMRI) signal in different brain regions of the Default Mode Network (DMN) and the Executive Control Network (ECN) at rest | Change from baseline functional network integrity at 12-weeks
  Resting state brain networks known to be vulnerable to decline with normal aging

SECONDARY OUTCOMES:
Motor learning rate | Change from baseline learning rate at 12-weeks
  Learning rate parameter expressing rate of reaction time speeding in an alternating serial reaction time task (ASRTT)
Explicit paired associates learning rate | Change from baseline learning rate at 12-weeks
  Learning rate parameter expressing rate of improvement in accuracy in a paired associates learning task
Executive function composite measure | Change from baseline executive function performance at 12-weeks
  Composite score from performance (speed and accuracy) on four executive function tasks, including Trails A and B, Go/No-Go dual task, a modified flanker task, and a non-verbal working memory n-back task
Cardiovascular fitness measured as "Vo2 max" from a cycle ergometer test | Change from baseline fitness at 12-weeks
  The ability of the heart and lungs to supply oxygen to working muscle tissues and the ability of the muscles to use oxygen to produce energy for movement

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Voss, PhD, Principal Investigator — University of Iowa
Locations (1):
- HBC Lab, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
In accord with NIH regulations, we will make the data and relevant documentation available to other investigators at their request upon acceptance of the main findings from the study for publication. Because the collected data are to remain anonymous, only a subject number will identify all data. To further protect the privacy and confidentiality of the data, data and documentation will be made available only under a data-sharing agreement that provides for restrictions for the transferring of data to others and a commitment that the data will be used for research purposes only and not for a profit-making enterprise.

REFERENCES:
- [Derived] Voss MW, Weng TB, Narayana-Kumanan K, Cole RC, Wharff C, Reist L, Dubose L, Sigurdsson G, Mills JA, Long JD, Magnotta VA, Pierce GL. Acute Exercise Effects Predict Training Change in Cognition and Connectivity. Med Sci Sports Exerc. 2020 Jan;52(1):131-140. doi: 10.1249/MSS.0000000000002115. PMID 31385912